CLINICAL TRIAL: NCT07241364
Title: Effect of the Superficial Cervical Plexus Block in the Hypotensive Anesthesia of Ear Surgery.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Lydia edward aziz zakhary, lecturer of anesthesia , intensive care and pain management, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: cervical plexus block
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Pain After Surgery
Keywords: cervical plexus block; hypotensive anesthesia; ear surgery
MeSH Terms: interventions — Nerve Block

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): will receive only conventional general anasthesia in ear surgery
- study group (Experimental): patients will receive superficial cervical plexus block in addittion to general anesthesia
  Interventions: Procedure: nerve block with bupivacaine 0.25%

INTERVENTIONS:
Procedure: nerve block with bupivacaine 0.25% — superficial cervical plexus block (superficial CPB ) will be administered in a supine position with the head turned opposite to the side of the block using ultrasound guidance .
  Local anaesthetic will be injected alongside the posterior border of the muscle 2-3 cm in cranial and caudal directions. Using a 'fan' technique, the local anaesthetic will be administered subcutaneously and behind the sternocleidomastoid muscle. Ten millilitres of 0.25% bupivacaine were injected for each side of the block using a 1.5-inch 24-gauge needle..
  Arms: study group

SUMMARY:
We aimed to evaluate the analgesic effect of ultrasound guided Superficial cervical plexux block in tympanomastoid ear surgeries by comparing it with conventional general anaesthesia using systemic analgesic through observation of intra- and postoperative requirements of the total dose of systemic analgesics, visual analog scale (VAS) score, total duration of analgesia, vital parameters and the occurrence of any perioperative complications.

DETAILED DESCRIPTION:
Patients meeting the inclusion criteria were randomly assigned into two groups, the control group and the study group, by a computer-generated randomization program. All patients in both group will be informed by the study methods,aim, side effect in clear language, written consent will be taken in clear spoken and written language, All patients of both groups ,once arrived to the OR, monitor will be attached, baseline SBP, DBP,MAP,SPO2,PULSE will be recorded, General anaesthesia (GA) will be induced with intravenous inj. of propofol 2-2.5 mg/kg, , fentanyl 1 microgram/kilogram (μg/kg). and atracuruim 0.5 mg/kg was given for muscle relaxation .

In study Group patients, superficial CPB will be administered in a supine position with the head turned opposite to the side of the block using ultrasound guidance .

Local anaesthetic will be injected alongside the posterior border of the muscle 2-3 cm in cranial and caudal directions. Using a 'fan' technique, the local anaesthetic will be administered subcutaneously and behind the sternocleidomastoid muscle. Ten millilitres of 0.25% bupivacaine were injected for each side of the block using a 1.5-inch 24-gauge needle. [2].

General anaesthesia will maintained with O2 + air (50:50), 3-litre flow, sevoflurane 2% to 2.5% and an intravenous inj. of atracuiruim 0.01 mg/kg every 20 min. An intraoperative rise in heart rate (>100/min) and systolic blood pressure (≥ 20% from pre-induction value) will be recorded and managed by giving intravenous inj. of fentanyl 0.5 microgram/kg in incremental doses (dose of fentanyl did not exceed 3 μg/kg for less than three hours of surgery). At the end of the surgery, the reversal of residual neuromuscular block will be done and the patient will be extubated. The patient will be then transferred to the recovery room and the severity of pain will be assessed by a VAS scale ( visual analog score scale ), which is a straight line denoting one end with no pain and the other end with the worst pain. VAS score was calculated as follows: 0, no pain; 1-3, mild pain; 4-6, moderate pain; 7-9, severe pain; 10, worst pain. The VAS score will be assessed when the patient could follow verbal commands.

Evaluation of block for adequate analgesia intraoperatively will be done in terms of the total requirement of intravenous analgesics through the observation of heart rate and blood pressure and postoperatively, it will be done by observing VAS score, time of first demand for a bolus of rescue analgesic (intravenous paracetamol) and total requirement of rescue analgesic in 24 hours.. Pulse, mean blood pressure (BP), oxygen saturation (SpO2) and any side effects were also noted.

ELIGIBILITY:
Inclusion Criteria:

1 - Both genders. 2- Age between 20 -40 years. 3- ASA 1 & 2 physical status. 4- Patients undergoing simple ear surgery as Tympano-mastoidectomy

Exclusion Criteria:

* 1- Infection at or near the injection site. 2- Uncontrolled preoperative hypertension. 3- age < 20 or >40 4- chronic opoid abuse patients. 5- patients with pre existing neuropathy or other neurological diseases. 6- patients on anticoagulation. 7- plt count < 100 or INR > 1.7 8- lengthy surgery more than 3 hours . 9- hypersensitivity to local anesthetics. 10- patients with psychiatric illness.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-11-20 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
pain | 24 hours
  monitoring pain score using visual analog score (VAS) postoperative . to evaluate the analgesic effect
analgesia | 24 hours
  The number of analgesic doses required for each patient as rescue analgesia (when VAS > 3), will be recorded and statistically compared between the two groups

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ho B, De Paoli M. Use of Ultrasound-Guided Superficial Cervical Plexus Block for Pain Management in the Emergency Department. J Emerg Med. 2018 Jul;55(1):87-95. doi: 10.1016/j.jemermed.2018.04.030. Epub 2018 May 29. PMID 29858144